CLINICAL TRIAL: NCT03776968
Title: A Study Evaluating HC-1119 Single-Dose Pharmacokinetics and Effect of Food on Its Pharmacokinetics in Healthy Chinese Adults
Brief Title: A Study Evaluating HC-1119 Single-Dose Pharmacokinetics and Effect of Food on Its Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC-1119-PK
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HC1119 (Experimental): Fasting state:40 mg, 80 mg, 160 mg; After meal: 160mg;
  Interventions: Drug: HC1119

INTERVENTIONS:
Drug: HC1119 — oral

SUMMARY:
This is a phase I study evaluating HC-1119 single-dose pharmacokinetics and effect of food on its pharmacokinetics in healthy Chinese adults. The study primary objective is to evaluate the HC-1119 pharmacokinetic characteristics and the effect of food on its pharmacokinetics in healthy Chinese males, subsequent to a single oral administration of HC-1119 with different doses in healthy Chinese males.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form.
2. Healthy Chinese male aged between 18-45 years old (inclusive).
3. Weight ≥ 50.0 kg, and BMI between 19.0-26.0 kg/m2 (inclusive) at screening. BMI = weight (kg) / height2 (m2).
4. Defined as "healthy" based on past medical history, physical examination, vital signs, laboratory tests, 12-Lead ECG, and chest x-ray performed at screening. All examination results must be within the normal range corresponding to the subject's age and gender, or determined by the investigator as "no clinical significance (NCS)" when the result is out of range.
5. All male subjects and their female spouses/sexual partners with child-bearing potential must adopt continuous and effective contraceptive methods, that is, two forms of contraception should be performed spontaneously (including at least one barrier method), from the initiation of screening and the whole study period to at least three months after administration.
6. Able to maintain a consistency of good communication with the investigators, and understand and comply with all the requirements of this study.

Exclusion Criteria:

1. A history of cardiovascular, lung, hepatic, renal, respiratory, nervous system, musculoskeletal, endocrine, or GI disease, or a history of other serious systemic diseases.
2. A clinically significant history of drug allergies or a history of specific allergic disease (asthma, urticaria, eczema dermatitis), especially being allergic to any ingredients of the study drug or formulation.
3. Suffered (within 1 week prior to the study) or currently suffering from febrile illness, symptomatic viral infection, bacterial infection (including upper respiratory tract infection), or fungal infection (except skin infection).
4. Administered any prescription drugs, Chinese herbal medicine, OTC drugs, or food supplements (including vitamins) within 4 weeks prior to the study.
5. Administered any inducers or inhibitors of hepatic drug metabolism within 1 month prior to the study (such as: inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, and omeprazole; inhibitors - antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, and antihistamines).
6. History of seizures within 12 months prior to the study, including any history of febrile seizures, loss of consciousness, or transient ischemic attack, and any condition that increases the risk of seizures (such as history of stroke, cerebral arteriovenous malformation, traumatic brain injury with coma requiring hospitalization, and lacunar infarct).
7. Recent history (in the past 3 years) and/or current medical history of autonomic dysfunction (such as recurrent syncope and palpitations).
8. History of medication abuse or a positive urine drug screen within 12 months prior to the study.
9. Smokers or those who smoked more than 10 cigarettes per day (or equivalent amounts of tobacco) within 3 months prior to the study, or those who are unable to stop smoking during the entire course of the study.
10. History of alcohol abuse or those with regular consumption of alcoholic beverages (daily consumption exceeding 14 units of alcohol, 1 unit = 360 ml of beer, 45 ml of 40% liquor, or 150 ml of wine) within 6 months prior to the study, or having a positive breath alcohol test result.
11. Donated or lost blood ≥ 400 ml of blood within 3 months prior to the study.
12. Received treatment with any investigational drug or participated in any clinical trial within 3 months prior to the study.
13. Requiring a special diet and unable to follow a standardized diet.
14. Overconsumption of tea, coffee, and/or caffeinated beverages daily (more than 8 cups, 1 cup = 250 ml).
15. Consumed grapefruit or product containing grapefruit (such as jam) within 1 week prior to receiving the investigational drug.
16. Positive HIV, HBsAg, HCV, or syphilis test result.
17. Cannot complete this study for any other reasons, or determined by the investigator to be unsuitable for this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to infinity (∞) (AUC0-∞) | From the first dose of the study drug to day 50
Area under the plasma concentration-time curve from time 0 to time t of the last measurable concentration(AUC0-t) | From the first dose of the study drug to day 50
Peak concentration (Cmax) | From the first dose of the study drug to day 50
Peak time (Tmax) | From the first dose of the study drug to day 50
Elimination half life (t1/2) | From the first dose of the study drug to day 50
Apparent clearance (CL/F) (prototype) | From the first dose of the study drug to day 50
Apparent volume of distribution (Vd/F) (prototype) | From the first dose of the study drug to day 50
Mean residence time (MRT) | From the first dose of the study drug to day 50

SECONDARY OUTCOMES:
Number of patients with adverse events | From the first dose of the study drug to day 50
  Safety measures

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital Ethics Committee, Shanghai, China

IPD SHARING:
Plan to Share IPD: No